CLINICAL TRIAL: NCT04453826
Title: A Multicenter Randomized Clinical Phase 3 Trial of Induction Chemotherapy Plus Concurrent Chemo-radiotherapy With or Without Camrelizumab for High Risk Nasopharyngeal Carcinoma
Brief Title: Concurrent and Adjuvant PD1 Treatment Combined With Chemo-radiotherapy for High-risk Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Yuebei People's Hospital (Other); Wuzhou Red Cross Hospital (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Chief Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-MYC-2020-1103
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Cancer; Chemotherapy; Radiotherapy; PD-1 Therapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab plus chemo-radiotherapy arm (Experimental): 3 cycles of gemcitabin and cisplatin induction chemotherapy plus concurrent chemo-radiotherapy with concurrent and adjuvant camrelizumab therapy.
  Interventions: Drug: Camrelizumab plus chemo-radiotherapy
- Chemo-radiotherapy arm (Active Comparator): 3 cycles of gemcitabin and cisplatin induction chemotherapy plus concurrent chemo-radiotherapy.
  Interventions: Drug: Chemo-radiotherapy alone

INTERVENTIONS:
Drug: Camrelizumab plus chemo-radiotherapy — 1. Camrelizumab: 200 mg, intravenous injection over 60 minutes (Q3W); 2 cycles of camrelizumab are concurrently used during radiotherapy and camrelizumab are maintained for 1 year after the end of radiotherapy.
  2. Gemcitabine plus cisplatin induction chemotherapy: gemcitabine is injected intravenously at the dose of 1000 mg/m2 on the 1st and 8th day (within 30 minutes) for 3 cycles; cisplatin is injected intravenously at the dose of 80 mg/m2 on the 1st day, for 3 cycles. 1 cycles per 3 weeks.
  3. Concurrent cisplatin chemotherapy: cisplatin is given at a dose of 100 mg/m2 via a continuous intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy for 2 cycles. 1 cycles per 3 weeks.
  4. IMRT: PTVnx#69.96Gy/33Fr/2.12Gy; PTVnd#69.96Gy/33Fr/2.12Gy; PTV1#59.4Gy/33Fr/1.8Gy; PTV2#54Gy/33Fr/1.64Gy
  Arms: Camrelizumab plus chemo-radiotherapy arm
Drug: Chemo-radiotherapy alone — 1. Gemcitabine plus cisplatin induction chemotherapy: gemcitabine is injected intravenously at the dose of 1000 mg/m2 on the 1st and 8th day (within 30 minutes) for 3 cycles; cisplatin is injected intravenously at the dose of 80 mg/m2 on the 1st day, for 3 cycles. 1 cycles per 3 weeks.
  2. Concurrent cisplatin chemotherapy: cisplatin is given at a dose of 100 mg/m2 via a continuous intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy for 2 cycles. 1 cycles per 3 weeks.
  3. IMRT: PTVnx#69.96Gy/33Fr/2.12Gy; PTVnd#69.96Gy/33Fr/2.12Gy; PTV1#59.4Gy/33Fr/1.8Gy; PTV2#54Gy/33Fr/1.64Gy
  Arms: Chemo-radiotherapy arm

SUMMARY:
Through multicenter, open-label, randomised clinical trials, we intend to demonstrate that concurrent and adjuvant PD-1 treatment added to chemo-radiotherapy could further decrease the rate of disease progression and improve the survival outcome of high risk patients with nasopharyngeal carcinoma compared with those treated with chemo-radiotherapy alone.

DETAILED DESCRIPTION:
Through multicenter, open-label, randomised clinical trials, high risk patients with nasopharyngeal carcinoma (staged as II-III with SD/PD according to RECIST criteria or EBV DNA of >0 copies/mL after 3 cycles of GP induction chemotherapy and staged as IVa) are randomized into camrelizumab plus chemo-radiotherapy arm and chemo-radiotherapy arm. The efficacy and safety of patients between these two arms are compared.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated type, i.e., WHO type II or type III).
2. Staged as T4N0-2M0,T1-4N3M0 (stage IVa) at diagnosis (according to the 8th AJCC edition).
3. Staged as T1-3N1-2M0, T2-3N0M0 (stage II-III) with SD/PD according to RECIST criteria or EBV DNA of >0 copies/mL after 3 cycles of GP induction chemotherapy.
4. Aged between 18-70 years.
5. Karnofsky scale (KPS)≥70.
6. Normal bone marrow function.
7. Normal liver and kidney function:

   1. total bilirubin, AST and ALT levels of no more than 2.5 times the upper normal limit;
   2. creatinine clearance rate of at least 60 mL/min or creatinine of no more than 1.5 times the upper normal limit.
8. Given written informed consent.

Exclusion Criteria:

1. Histologically confirmed keratinized squamous cell carcinoma (WHO type I) or basal squamous cell carcinoma.
2. Recurrent or metastatic nasopharyngeal carcinoma.
3. Staged as II-III which is evaluated as PR or CR and EBV DNA of 0 copies/mL after 3 cycles of GP induction chemotherapy.
4. Has known allergy to large molecule protein products or any compound of study therapy.
5. Has known subjects with other malignant tumors.
6. Has any active autoimmune disease or history of autoimmune disease.
7. Has a history of psychiatric substance abuse, alcoholism, or drug addiction.
8. The laboratory examination value does not meet the relevant standards within 7 days before enrollment
9. Received a systematic glucocorticoid therapy within 4 weeks of the first dose of study medication.
10. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB with 1 year.
11. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent.
12. Has active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy). Patients with skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) will be allowed to enroll.
13. Has a known history of human immunodeficiency virus (HIV).
14. Has hepatitis B surface antigen (HBsAg) positive with HBV DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.
15. Has received a live vaccine within 4 weeks of planned start of study therapy.
16. Pregnancy or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomisation to the date of first distant metastases.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Incidence of treatment related acute complications | up to 1 years
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
Incidence of treatment related late complications | up to 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | up to 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | up to 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

REFERENCES:
- [Derived] You R, Xu GQ, Ding X, Liang JH, Liu ZG, Zou X, Liu YP, Hu GY, Liu YM, Duan CY, Liu LZ, Zhang WJ, Liu Q, Li HF, Ouyang YF, Duan XT, Wang Q, Peng L, Liang JL, Feng ZK, Qin ZH, Liu X, He ZK, Zhang B, Long GX, Jiang YH, Lei F, Huang PY, Hua YJ, Chen MY. Standard chemoradiotherapy with concurrent and adjuvant camrelizumab in patients with high risk nasopharyngeal carcinoma: multicentre, randomised, open label, phase 3 trial. BMJ. 2026 Feb 10;392:e085863. doi: 10.1136/bmj-2025-085863. PMID 41667193